CLINICAL TRIAL: NCT04404309
Title: Patient Characteristics, Validity of Clinical Diagnoses and Outcomes Associated With Suicidality in Inpatients With Symptoms of Depression (OASIS-D)
Brief Title: Outcomes Associated With Suicidality in Inpatients With Symptoms of Depression (OASIS-D)
Acronym: OASIS-D
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Principal Investigator, Prof. Dr. med Christoph Correll, Clinic Director, Charite University, Berlin, Germany
Other Study IDs: EA2/061/20
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Depression; Depression Moderate; Depression Severe; Suicidal and Self-injurious Behavior; Suicidal Ideation; Suicide, Attempted
Keywords: Depression; Suicidality
MeSH Terms: conditions — Depression; Self-Injurious Behavior; Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Population 1: Any patient admitted to a psychiatric ward with a clinical diagnosis of (unipolar) major depression
- Population 2: Any patient with a clinical diagnosis of a moderate or severe unipolar depressive disorder with suicidal tendencies that persist for at least 48 hours after admission
- Population 3: Patients with moderate or severe unipolar depressive episodes validated by research interviews and suicidal tendencies that persist for at least 48 hours after admission who will be followed up for 6 months

SUMMARY:
This 6-month, naturalistic cohort study examines male and female inpatients aged 18 to 75 years i) with any form of unipolar depressive episode (cohort 1); ii) clinical diagnosis of a moderate or severe unipolar depressive episode and suicidal tendencies who agree to participate in a prospective study (cohort 2); and moderate or severe unipolar depressive episodes validated by research interviews and and suicidal tendencies that persist for at least 48 hours after admission who are followed up for 6 months (cohort 3).

DETAILED DESCRIPTION:
Epidemiological cross-sectional study in over 3000 inpatients with a clinical diagnosis of major depressive disorder, validation of the clinical diagnosis in 520 patients, and prospective naturalistic 6-month follow-up study of 260 adults with a research interview-confirmed major depressive disorder, with data collection at the following points: at T0 = time of hospitalization (epidemiological study population 1 with data from clinical routine practice), at time T1 of baseline survey in patients with persistent suicidal tendencies, i.e. at least 48 hours after T0 (study population 2 as a subgroup of study population 1, with study information and consent), and in study population 3 (subgroup of study population 2, with study information and consent) at the time of discharge (T2), 3 months after admission to hospital (T3/ by telephone) and 6 months after inpatient admission (T4).

The aim of the study is to characterize the remission or recurrence of suicidal symptoms in the context of a depressive episode. It is expected that the results will help to improve the understanding of the disease process and the further development of effective intervention options.

ELIGIBILITY:
Inclusion Criteria:

For Population 1

1.any form of unipolar depressive episode

For Population 2

1. clinical diagnosis of a moderate or severe unipolar depressive episode
2. clinically diagnosed suicidal tendencies that persist for at least 48 hours after admission to hospital
3. Written consent to participate in the study

For Population 3

1. Diagnosis of a moderate or severe unipolar depressive disorder through the structured research interview "Mini International Neuropsychiatric Interview" (M.I.N.I.)
2. Suicidality with a value > / = 1 for item 2 (passive suicidality) OR item 3 (active suicidality) based on the research interview "Sheehan Suicidality Tracking Scale" (S-STS)
3. Written consent to participate in the study

Exclusion Criteria:

* Patients younger than 18 years or older than 75 years
* No clinical diagnosis of a depressive episode
* Depressive episode in the context of a bipolar disorder- secondary depression as a result of physical illness or substance use
* severe physical symptoms of disease that make participation in the study impossible
* Pregnancy
* not being able to understand the study processes
* incapable of giving informed consent
* no authorization to give consent due to (limited) incapacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient are gonna be recruited from 7 different psychiatric clinics. For population 1, only clinically available data is extracted from patient records population 2 and 3: Patients who meet the inclusion criteria and are in psychiatric hospital treatment in the study centres
Sampling Method: Non-Probability Sample
Enrollment: 3331 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sheehan Suicidality Tracking Scale (S-STS) | 20 min
  Interview for Suicidality, Suicidal Behavior and Suicide Attempts, the higher the value the worse the outcome, the values can range from 0- 156
Mini-International Neuropsychiatric Interview (M.I.N.I.) | 40 min
  Semi-structured interview for research diagnosis

SECONDARY OUTCOMES:
Clinical Global Impression of Resolution Suicide Risk (CGI-SR-R) | 1 min
  One Question rated by an interviewer
Clinical Global Impression of Imminent Suicide Risk (CGI-SR-I) | 1 min
  One Question rated by an interviewer
Clinical Global Impression - Severity (CGI-S) | 1 min
  One Question about severity of illness, rated by an interviewer
Clinical Global Impression - Change (CGI-C) | 1 min
  One Question about change of the symptoms rated by an interviewer
Young Mania Rating Scale (YMRS) | 20 min
  Structured Interview for Mania Symptoms
Montgomery-Asberg Depression Rating Scale (MADRS) | 20 min
  Structured Interview for Symptoms of Depression
Service Use and Resource Form (SURF) | 30 min
  Structured Interview for Service Use of the health care system
Adherence Questions | 5 min
  Semi Structured Interview for Adherence of Antipsychotics

CONTACTS AND LOCATIONS:
Overall Officials: Christoph U Correll, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité, Mitte, Germany

REFERENCES:
- [Derived] Nohles VB, Bermpohl F, Schoofs N, Bathe-Peters R, Hilpert N, Dafsari FS, Reif-Leonhard C, Reif A, Schillo S, Arshad RS, Getty P, Falkai P, Schule C, Wang E, Adli M, Papenfuss R, Meyer-Lindenberg A, Fritze S, Otte C, Piber D, Graumann L, Weyn-Banningh S, Bauer M, Lewitzka U, Spreer M, Clemens J, Rubarth K, Correll CU. Clinical and Treatment Characteristics of 3795 Adults Consecutively Hospitalized for Major Depressive Disorder in the OASIS-D Study. Depress Anxiety. 2025 Nov 26;2025:4470169. doi: 10.1155/da/4470169. eCollection 2025. PMID 41347111
- [Derived] Nohles VB, Bermpohl F, Falkai P, Reif-Leonhard C, Jessen F, Adli M, Otte C, Meyer-Lindenberg A, Bauer M, Rubarth K, Anghelescu IG, Rujescu D, Correll CU. Patient characteristics, validity of clinical diagnoses and Outcomes Associated with Suicidality in Inpatients with Symptoms of Depression (OASIS-D): design, procedures and outcomes. BMC Psychiatry. 2023 Oct 13;23(1):744. doi: 10.1186/s12888-023-05230-9. PMID 37828493